CLINICAL TRIAL: NCT06726941
Title: Effect of Exercise on Neuroplasticity-Related Gene Expression and Histone Modifications in Patients With Hemiplegia
Brief Title: Effect of Exercise Gene Expression and Histone Modifications in Patients With Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Hasan Toktaş, Professor, Afyonkarahisar Health Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBBEPIGENETIC
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke, Acute; Acute Hemiparesis
Keywords: ischemic stroke; acute hemiplegia; epigenetics
MeSH Terms: conditions — Ischemic Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: All participants enrolled will receive the same treatment. Gene analysis, histone acetylation levels, motor function and quality of life changes will be assessed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): This group consists of post-stroke hemiplegia participants who will be included in a physiotherapy and rehabilitation program to evaluate the effects on neuroplasticity-related gene expression and histone modification levels, spasticity levels, motor functions, daily living activities, and quality of life.
  Interventions: Other: Physiotherapy and Rehabilitation Practices

INTERVENTIONS:
Other: Physiotherapy and Rehabilitation Practices — It was planned to give the participants a routine stroke rehabilitation program consisting of 45 minutes of active, passive range of motion exercises and strengthening exercises, balance exercises, walking training and 20 minutes of bicycle ergometry, accompanied by a physiotherapist with at least 5 years of experience in stroke rehabilitation. It was planned to give passive bicycle ergometry to patients without voluntary muscle movement and muscle strength, and active bicycle ergometry to participants with voluntary muscle movement and muscle strength, with the bicycle rehabilitation. It was planned to apply the exercise program to the patients for 5 days a week and for a total of 30 sessions. It will be recommended that they continue the medical treatment they are using during the treatment program. Routine evaluations will be made by the physiatrist before the rehabilitation program starts and 2 tubes of venous blood will be taken from the patients by an experienced nurse

SUMMARY:
The aim of this study is to demonstrate the effect of routine exercise program on neuroplasticity through histone acetylation and gene expression changes in acute stroke survivors from an epigenetic perspective and to investigate the correlation of epigenetic effects with its effects on motor function and quality of life.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of disability worldwide. Hemiplegia is the name of the clinical condition that occurs after a stroke. It is the loss of strength in the arm, leg and sometimes the face on one side of the body. Rehabilitation is vital to minimize the sequelae after a stroke, and patients who undergo continuous professional and systematic rehabilitation after the acute phase tend to recover rapidly. An important therapeutic goal of motor recovery is to maximize neuronal plasticity and facilitate motor tasks through motor learning during therapeutic exercise in the neurorehabilitation of patients with motor dysfunction. In particular, intact motor-related regions of the brain are expected to compensate for the impaired neuronal systems. Therefore, therapeutic exercise is expected to compensate for the impaired neuronal system by altering the (cortical) neuronal network as well as the expression of postsynaptic receptors, presynaptic neurotransmitters, regeneration, modulation and synaptic formation at cortical synapses. Epigenetic mechanisms regulate gene transcription based on modifications of DNA promoter regions and histones in chromatin. Epigenetic mechanisms include various DNA and histone modifications (i.e., methylation and acetylation of DNA and histones). In particular, the acetylation level of specific lysine residues in histones is one of the most powerful epigenetic modifications and is essential for transcriptional regulation. Studies show that exercise reduces the expression and activity of HDACs and increases histone acetylation, upregulating the expression of genes important for neuroplasticity.

Some genes associated with neuroplasticity are:Brain-Derived Neurotrophic Factor (BDNF) , Cyclic adenosine monophasphate Response Element-Binding Protein (CREB1), Growth Associated Protein 43 (GAP43), Neurotrophic Receptor Tyrosine Kinase 2 (NTRK2), Synapsin I (SYN1).

Histone H3 Lysine 27 Acetylation (H3K27ac) plays a critical role in the epigenetic regulation of gene expression and is associated with processes such as neuroplasticity, memory, and learning. Various studies have shown that environmental factors such as exercise can increase H3K27ac levels and thus support neuroplasticity.

In this study, participants with acute hemiplegia will be given the same routine rehabilitation program. Neuroplasticity-related gene expression and histone acetylation levels will be compared in venous blood taken from the patient before and after exercise.

In addition, the patient will be examined before and after exercise, and routine Mini-Mental Test, Brunnstrom, Fulg-Meyer upper and lower extremity evaluation, Spasticity evaluation with modified ashworth scale, Functional Independence Scale, ABILHAND Stroke Hand Function Questionnaire, Stroke Impact Questionnaire, 10-meter walking test will be performed to evaluate quality of life and motor function.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who applied to Afyonkarahisar Health Sciences University Physical Therapy and Rehabilitation Clinic for rehabilitation purposes and had a stroke for the first time
2. Participants with ischemia as the etiology of stroke
3. Participants between the ages of 25-70
4. Drugs that have been used for at least 1 month and up to 6 months after a cerebrovascular accident

Exclusion Criteria:

1. Participants whose stroke etiology is other than ischemia
2. Participants with clinically significant neurological disease other than stroke
3. Participants with systemic and musculoskeletal diseases that will not tolerate neurological rehabilitation and prevent them from participating

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Genetic analyses | Baseline (pre-treatment) and 6 weeks (post-treatment)
  Real-Time Polymerase Chain Reaction (PCR) method will be used to determine the expression of BDNF, CREB1, GAP43, NTRK2 and SYN1 genes from the peripheral venous blood samples of the participants. The region of interest will be amplified in the Real-Time PCR device using primer pairs specific to the relevant genes. Changes in gene expressions in patients before and after treatment will be determined.
Histone Proteins | Baseline (pre-treatment) and 6 weeks (post-treatment)
  Leukocytes will be isolated from blood samples before and after exercise. Isolation of histone proteins will be performed from the isolated leukocytes using the relevant isolation procedures. Pre- and post-treatment levels will be compared.
Histone Acetylation Analysis | Baseline (pre-treatment) and 6 weeks (post-treatment)
  H3K27ac levels in the isolated histone proteins will be determined colorimetrically based on the ELISA method. Pre- and post-treatment levels will be compared.

SECONDARY OUTCOMES:
Neurophysiological Assessment | Baseline (pre-treatment) and 6 weeks (post-treatment)
  Brunnstrom Staging is a test that evaluates the motor development of hemiplegic patients. In this test, the neurophysiological recovery process of hemiplegic patients is defined as 6 stages. According to this staging, the lowest stage is stage 1 (flaccid, no voluntary movement stage), and the highest stage is stage 6 (isolated joint movement stage). In Brunnstrom staging, the hand, upper extremity and lower extremity are evaluated separately.
Spasticity Assessment | Baseline (pre-treatment) and 6 weeks (post-treatment)
  Spasticity was planned to be evaluated with the Modified Ashworth Scale (MAS). In MAS, patients are evaluated over 5 points. 0 indicates no increase in muscle tone, and 4 indicates that the extremity is rigid in the flexion and extension directions.
Functional independence scale (FIM) | Baseline (pre-treatment) and 6 weeks (post-treatment)
  It is a widely applied, validated and reliable approach to functional assessment in Turkish society. FIM analyzes two different aspects of disability, namely motor and cognitive functions. FIM is a scale consisting of 6 subgroups, namely self-care (42 points), sphincter control (14 points), transfer (21 points), movement (14 points), communication (14 points) and social perception (21 points), and evaluates 18 activities. Each activity is evaluated in terms of functional independence using a 7-point scale. Higher scores indicates independence.
Fugl Meyer Upper Extremity Evaluation Questionnaire | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The Fugl-Meyer Upper Extremity Motor Evaluation Questionnaire (FMUE Questionnaire) was developed to quantitatively assess sensorimotor recovery after stroke. It was prepared based on Brunnstrom's stages of motor recovery. The FMUE Questionnaire consists of 33 items, each scored from 0 to 2, where 0 = cannot perform, 1 = partially performs, and 2 = fully performs. The total score is 66. A range of data is available for the FMUE Questionnaire for clinically important minimum differences. A change of 4 to 7 points in chronic stroke and 9 to 10 points in subacute stroke is considered clinically significant.
A Rasch-built measure of manual ability(ABILHAND) Stroke Hand Function Questionnaire | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The ABILHAND Hand Questionnaire was developed in 1998 to measure patient-perceived hand dexterity. It contains 23 questions regarding the patient's difficulty in performing activities. One of the following options is marked: impossible (0 points), difficult (1 point), easy (2 points). The total score is 46.
Stroke Impact Questionnaire | Baseline (pre-treatment) and 6 weeks (post-treatment)
  Stroke Impact Scale (SIS) is a stroke-specific health status measure. It consists of 59 items and 8 sections. The patient is asked to evaluate the difficulty experienced in completing each item in the last week on a five-point Likert scale. One point indicates that the patient could not complete the item, and five points indicate that he/she had no difficulty in completing it. It also includes a visual analog scale (0: No improvement, 100: Full recovery) regarding the general perception of recovery after stroke. A Turkish validity and reliability study has been conducted.
10 meter walk test | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The 10 Meter Walk Test is a performance measure used to assess walking or walking speed in meters per second over a short distance. It can be used to determine functional mobility, gait and vestibular function. Participants are asked to walk at maximal speed for 14 m. Marks are placed on the floor for a 2 m acceleration and a 2 m deceleration, a starting point and an ending point. Measurement is started at 2 m. Measurement is finished at 12 m. The time taken for the walk is measured manually using an electronic timer for all participants. The total time for the 10 meter walk is recorded. The 10 m is then divided by the total time (in seconds) taken to complete it. The total time is recorded in m/s. Shorter time duration means better mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Toktas, Professor, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] Xing Y, Bai Y. A Review of Exercise-Induced Neuroplasticity in Ischemic Stroke: Pathology and Mechanisms. Mol Neurobiol. 2020 Oct;57(10):4218-4231. doi: 10.1007/s12035-020-02021-1. Epub 2020 Jul 20. PMID 32691303
- [Background] Maejima H, Kitahara M, Takamatsu Y, Mani H, Inoue T. Effects of exercise and pharmacological inhibition of histone deacetylases (HDACs) on epigenetic regulations and gene expressions crucial for neuronal plasticity in the motor cortex. Brain Res. 2021 Jan 15;1751:147191. doi: 10.1016/j.brainres.2020.147191. Epub 2020 Nov 2. PMID 33152341
- [Background] Penna LG, Pinheiro JP, Ramalho SHR, Ribeiro CF. Effects of aerobic physical exercise on neuroplasticity after stroke: systematic review. Arq Neuropsiquiatr. 2021 Sep;79(9):832-843. doi: 10.1590/0004-282X-ANP-2020-0551. PMID 34669820
- See also: A Review of Exercise-Induced Neuroplasticity in Ischemic Stroke. — http://pubmed.ncbi.nlm.nih.gov/32691303/
- See also: Effects of exercise and pharmacological inhibition of histone deacetylases (HDACs) on epigenetic regulations and gene expressions crucial for neuronal plasticity in the motor cortex. — http://pubmed.ncbi.nlm.nih.gov/33152341/
- See also: Effects of aerobic physical exercise on neuroplasticity after stroke. — http://pubmed.ncbi.nlm.nih.gov/34669820/